CLINICAL TRIAL: NCT02901145
Title: A Phase I/II Clinical Trial of Nivolumab in Progressive/Relapsed Pediatric Solid Tumors
Brief Title: Nivolumab in Relapsed Pediatric Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0506-15-HMO
Record Dates: First submitted 2016-09-11; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Antibodies, Neoplasm
Keywords: immunotherapy,solid tumor,pediatric
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- progressive/relapsed solid tumors (Experimental): patient with progressive/relapsed solid tumors who failed first line therapy
  Interventions: Drug: Nivolumab,low dose cyclophosphamide

INTERVENTIONS:
Drug: Nivolumab,low dose cyclophosphamide — treatment with IV Nivolumab 3mg/kg every 2 weeks . after a month-addition of low dose cyclophosphamide at a starting dose of 50 mg/kg/day x7 days every 14 days with dose adaptation based on level of Tregulatory cells on follow up immunophenotype.

SUMMARY:
patients with progressive/relapsed solid tumors who failed first line therapy , will be treated biweekly with the anti PD1- Nivolumab. at least one month after treatment initiation low dose cyclophosphamide will be started .

patients on trial will submit tissue and blood tests for whole exome an immune genomic signature. patients will also undergo repeated immunophenotype as part of follow up.

DETAILED DESCRIPTION:
Programmed cell death 1 (PD-1) is an inhibitory receptor that prevents immune activation. PD-1 blockade can mediate reactivation of immune mediated tumor killing leading to tumor regression . Another mechanism of tumor associated immune inactivation is elevation of rates of T regulatory cells. This process may be prevented by treatment with low dose cyclophosphamide.

Objective:

This study will evaluate safety and tolerability of the anti PD1 antibody Nivolumab combined with other immunomodulating treatments, in pediatric patients with relapsed/progressive solid tumors

Method:

Patients will be treated with IV Nivolumab 3mg/kg over 60 minutes on day 1 and 15 of each cycle of 28 days.

1. Dose finding phase:

   1. Six patients will be accrued for the first cohort and treated for 1 month
   2. If an adverse event >grade 2 will occur in>2 patients, study medication dose will be reduced by 25% and another cohort of 6 patients will be accrued on the reduced dose.
   3. Dose finding cohorts will be accrued until determination of a dose with allowed DLT
2. Expansion phase

   1. Following dose determination patients will be accrued, to the final number of 30 patients
   2. Cyclophosphamide at the dose of 50 mg/dayx7days every 14 days (one week on one week off ) will be started . immunophenotype will be done every 28 days and dose of cyclophosphamide will be elevated by 25mg /day every month until highest ratio of CD8/CD25FOXP3 cells will be reached for every child
   3. All patients will be treated for 1 year or until imaging proven disease progression.
3. Required follow up

   1. All patients will undergo tumor bed imaging (CT/MRI-based on tumor location) with metastatic evaluation (according to standar follow up) every 4 months
   2. Tumor response will be measured based on RECIST criteria
   3. Toxicity assessment will be done according to the CTCAE v. 4.03

c. Collateral studies:

1. Immunohistochemical analysis for PD1 and PDL1 will be done on pretreatment paraffin embedded tissue to estimate it's ability to predict response.
2. Immune profile of peripheral blood lymphocytes including CD3+, CD4+, CD8+ FOX P3+ cells and it's correlation to objective response to therapy.
3. Exome sequencing of the tumor and peripheral blood will be done for every patient.

Exome will be evaluated for driver mutations and immunologic genomic signature.

ELIGIBILITY:
Inclusion Criteria:

1. Ages Eligible for Study: 12 Months and older
2. Patients must have had histologic verification of malignancy at original diagnosis or relapse

   Eligible pathologies:
   1. neuroblastoma following lack of complete response to at least two lines of therapy
   2. rhabdomyosarcoma following progression after first line therapy
   3. Ewing sarcoma following progression after second line of therpy
   4. Osteosarcoma following progression after first line of therapy all other pathologies will be discussed with PI
3. Patients must have measurable disease
4. Patient's current disease state must be one for which there is no known curative therapy
5. Karnofsky >= 50 for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
6. Patients must have fully recovered from the acute toxic effects of all prior anti-cancer treatment

   1. At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
   2. At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
   3. at least 56 days must have elapsed after transplant or stem cell infusion; patients with prior allogeneic transplants are not eligible
7. Blood counts recovery including ANC >= 750/mm^3 and Platelet count >= 50,000/mm^3
8. Creatinine clearance ≤ 1.5 ULN
9. liver function:Total bilirubin ≤ 2 ULN, ALT or AST ≤ 2.5 ULN (or < 5 in case of liver impairment)
10. Life expectancy of at least 4 months
11. Pregnancy:

    1. Negative pregnancy test in women of childbearing potential
    2. Use of an effective contraceptive method during the whole treatment and
    3. up to 3 months after the completion of treatment in males and females
12. prior informed consent signed

Exclusion Criteria:

1. Patients requiring daily systemic corticosteroids are not eligible; patients must not have received systemic corticosteroids within 7 days of enrollment on study
2. Patients who are currently receiving another investigational drug are not eligible
3. Patients who are currently receiving other anti-cancer agents are not eligible
4. Patients with a history of any grade autoimmune disorder are not eligible; asymptomatic laboratory abnormalities (e.g. antinuclear antibody [ANA], rheumatoid factor, altered thyroid function studies) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder
5. Patients with >= grade 2 hypothyroidism due to history of autoimmunity are not eligible; note: hypothyroidism due to previous irradiation on thyroidectomy will not impact eligibility
6. Patients who have an uncontrolled infection are not eligible.
7. Patients with active autoimmune disease. (any autoimmune state requiring medical treatment-including chronic medications)all immune modifying drugs should be stopped at least 7 days prior to enrollment.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 6 months
  Rate of patients with stable disease/tumor response at 6 months
Overall survival | 6 and 12 months
  Rate of patients alive at 6 months and 12 months

SECONDARY OUTCOMES:
evaluation of predictors for response | 12 months
  correlation between levels of PD1 receptor expression in the tumor and genomic signature with response

IPD SHARING:
Plan to Share IPD: No